CLINICAL TRIAL: NCT05242796
Title: Placebo Controlled, Randomized, Double Blind, Clinical Trial of the Effects of Low Frequency Magnet Therapy on Spasticity in Patients With Cerebral Palsy
Brief Title: Effects of Low Frequency Magnet Therapy on Spasticity in Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Armed Forces Hospital (Other Government)
Collaborators: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Ali AlGhamdi, Sr. Physical Therapy Specialist, King Fahad Armed Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFMMC
Record Dates: First submitted 2022-01-08; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12 sessions of magnet (Experimental)
  Interventions: Device: Low frequency magnetic therapy
- 24 sessions of magnet (Experimental)
  Interventions: Device: Low frequency magnetic therapy
- Placebo magnet intervention (Placebo Comparator)
  Interventions: Device: Low frequency magnetic therapy

INTERVENTIONS:
Device: Low frequency magnetic therapy

SUMMARY:
Background: Spasticity is a major challenge in patients with cerebral palsy (CP). It may cause unwanted complications and may affect the patient's quality of life. Currently there is no satisfactory long lasting control of spasticity. Many lines of evidence indicate that magnet therapy may be a useful intervention in the management of spasticity. Several studies showed that magnet may inhibit neuronal firing in the human nervous system; however, its effects weren't studied on spasticity. Objectives: The goal of the present study was to determine the short-and long-term effects of pulsed low frequency magnetic field therapy on spasticity in patient with CP. Methods: 48 patients with CP, who have measureable level of spasticity, were selected. The sample was divided randomly into active magnet group (received magnet therapy, 32 subjects) and placebo group (16 subjects). At the end of the 4th week the magnet group was divided into two sub-groups: 1st sub-group received magnet therapy for another 4 weeks while the other received the placebo. Measurements was taken at baseline, 4th, 8th and 12th weeks. Modified Ashworth Scale was used to measure spasticity, foot pressure platform system was used to measure the contact area and the maximum force of the feet, gross motor function measure (GMFM) was used to measure the functional level of the patients. The cerebral palsy quality of life (CP-QoL) questionnaire was used to measure the patients' various dimensions of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of diplegic or quadriplegic CP of both genders,
* Able to stand without assistance.
* Age from 4-16 years
* Measureable spasticity (1 or more according to the Modified Ashworth Scale).

Exclusion Criteria:

* Have recent organ transplants.
* Have heart pace maker.
* Have cardiac arrhythmia, tachy cardiac conditions or large aneurysm.
* Have heavy psychosis.
* Underwent any neuromuscular blockers of Spasticity.
* Underwent any surgery of tendon lengthening before or during the study.
* Have epileptic episodes.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Modified Ashowreth Scale at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  measure the muscle resistance following a passive stretch - grades from (0 - 4), lower score means better outcome
Change from baseline Gross Motor Function Scale at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  to evaluate the children with CP according to their motor functional ability - Scores (0% - 100%) where higher grade means better outcome.
Change from baseline Feet Contact Area at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  The weight distribution between the feet and the ground - Higher grade means better outcome
Change from baseline Feet Maximum Force at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  Measuring Feet Maximum Force of the participants - Higher grade means better outcome
Change from baseline Cerebral Palsy Quality of Live Questionnaire (Social well-being and acceptance dimension) at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (1,3,4,5,6,7,10,11,12,13,14,15).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome
Change from baseline Cerebral Palsy Quality of Live Questionnaire (Functioning dimension) at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (8,22,23,24,27,29,34,35,37,38,39,40).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome
Change from baseline Cerebral Palsy Quality of Live Questionnaire (Participation and physical health dimension) at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (9,16,17,18,19,20,21,25,26,30,37).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome
Change from baseline Cerebral Palsy Quality of Live Questionnaire (Emotional well-being dimension) at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (2,28,31,32,33,52).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome.
Change from baseline Cerebral Palsy Quality of Live Questionnaire (Access to services dimension) at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (41, 42, 43, 53, 54, 55, 56, 57, 58, 59, 60, 61).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome.
Change from baseline Cerebral Palsy Quality of Live Questionnaire (Pain and impact of disability dimension) at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (44, 45, 46, 47, 48, 49, 50, 51).
  2. Each item has an answer from one to nine; where (1= not bothered at all) to (9 = very bothered).
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means worse outcome.
Change from baseline Cerebral Palsy Quality of Live Questionnaire (Family health dimension) at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (62, 63, 64, 65).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome.
Comparison of Modified Ashowreth Scale scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  measure the muscle resistance following a passive stretch - grades from (0 - 4), lower score means better outcome
Comparison of Gross Motor Function Scale scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  to evaluate the children with CP according to their motor functional ability - Scores (0% - 100%) where higher grade means better outcome.
Comparison of Feet Contact Area scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  The weight distribution between the feet and the ground - Higher grade means better outcome
Comparison of Feet Maximum Force scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  Measuring Feet Maximum Force of the participants - Higher grade means better outcome
Comparison of Cerebral Palsy Quality of Live Questionnaire (Social well-being and acceptance dimension) scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (1,3,4,5,6,7,10,11,12,13,14,15).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome
Comparison of Cerebral Palsy Quality of Live Questionnaire (Functioning dimension) scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (8,22,23,24,27,29,34,35,37,38,39,40).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome
Comparison of Cerebral Palsy Quality of Live Questionnaire (Participation and physical health dimension) scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (9,16,17,18,19,20,21,25,26,30,37).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome
Comparison of Cerebral Palsy Quality of Live Questionnaire (Emotional well-being dimension) scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (2,28,31,32,33,52).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome.
Comparison of Cerebral Palsy Quality of Live Questionnaire (Access to services dimension) scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (41, 42, 43, 53, 54, 55, 56, 57, 58, 59, 60, 61).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome.
Comparison of Cerebral Palsy Quality of Live Questionnaire (Pain and impact of disability dimension) scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (44, 45, 46, 47, 48, 49, 50, 51).
  2. Each item has an answer from one to nine; where (1= not bothered at all) to (9 = very bothered).
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means worse outcome.
Comparison of Cerebral Palsy Quality of Live Questionnaire (Family health dimension) scores between the three groups from baseline at 4, 8 and 12 weeks | baseline, 4th week, 8th week and 12th week
  1. Items numbers in the questionnaire: (62, 63, 64, 65).
  2. Each item has an answer from one to nine; where 1= very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.
  3. To be calculated by summation of all the dimension's score.
  4. Higher score means better outcome.